CLINICAL TRIAL: NCT07364643
Title: Assessment of Asthma Management in Children Over 6 Years of Age and Their Caregivers. Implications for the Implementation of the SMART Strategy in Pediatrics.
Brief Title: Effectiveness of an Educational Intervention on Asthmatic Children in Inhaled Technique and Adherence.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Victòria Morón Faura, Principal Investigator, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-EMA-2025-05
Record Dates: First submitted 2025-09-22; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Asthma Childhood
Keywords: inhaler technique; treatment adherence; asthma self-management; nursing intervention
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population will be pediatric patients with a diagnosis of asthma, scheduled for consultation (Experimental): The included population will undergo an objective assessment with pulmonary function tests and will be given questionnaires to evaluate their knowledge about asthma treatment. Afterwards, they will receive a brief educational intervention and will be scheduled for a follow-up visit at 6 months to reassess pulmonary function parameters and knowledge level.
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Educational Intervention:
  The nurse will deliver a brief health education session focused on:
  1. Understanding the treatment. Provide clear information adapted to the patient's level, supported with visual aids.
  2. Distinguishing between maintenance and rescue treatment. Explain the role of each medication with practical examples.
  3. Assessment and correction of inhaler technique. Carry out a step-by-step demonstration and ask the patient to repeat the technique. Use educational materials (placebo devices, videos, diagrams) and reinforce learning with the teach-back method.
  4. Promoting autonomy. Encourage the patient to take part in administering the medication and foster self-management of the device.
  5. Evaluating and improving adherence. Suggest daily routines, reminders, and the use of alarms or mobile apps.
  6. Appropriate use of rescue medication. Involve the patient in decision-making, promote self-observation, and provide a clear action plan.

SUMMARY:
The goal of this study is to see if a short educational session and demonstration by a nurse can help asthmatic children (6-17 years-old), under hospital control, to manage their asthma better, to use their inhaler correctly, and to know when it should be used.

The main question it aims to answer is how much improvement is reached on asthma self-management. The comparison group is the same group. Researchers will compare results before and after educational intervention.

DETAILED DESCRIPTION:
The goal of this study is to see if a short educational session and demonstration by a nurse can help children manage their asthma better, use their inhaler correctly, and know when it should be used.

The study lasts about six months and has two visits:

Visit 1:

Participants will do the usual breathing tests, will show the nurse how to use the inhaler, and answer a few short questionnaires.

Then, the nurse will give some practical education using pictures and demonstrations. She will explain the right way to use the inhaler, to know the device, go over when and why to use inhaled medicine, and teach the participant how to recognize when asthma is getting worse and what can participant do about it.

Visit 2 (after 6 months):

Participants will repeat the same breathing tests and answer questionnaires again, so investigators can see what has changed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma.
* Prescribed treatment with inhaled corticosteroid.
* First-degree relative of the patient.

Exclusion Criteria:

. Inability to understand Spanish.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 428 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Correct inhaler technique | From the nursing intervention until the following 6 months.
  For the qualitative variable "inhaler technique," the Inhaler Technique Questionnaire (InTeQ), validated in pediatrics for the use of pressurized inhalers, will be used. This questionnaire includes 5 items considered critical, with an additional item, "shake the device," added for those using pMDIs.
  The 5 critical steps assessed are: exhale completely before inhalation, close lips firmly, inhale deeply, hold breath afterward, and exhale slowly, which are applicable to both pressurized metered-dose inhalers (pMDI) with a spacer and dry powder inhalers (DPI). The item "device activation" was removed, as it is inherent to the procedure and to facilitate practical applicability.

SECONDARY OUTCOMES:
Change in Treatment Adherence | From the nursing intervention until the following 6 months.
  It will be used the only specific questionnaire designed to measure adherence to inhalers, called the Inhaler Adherence Test (IAT). It consists of 10 items to be completed by the patient/caregiver when we want to identify patients with low adherence, and 2 additional items to be completed by the healthcare professional, which are specifically intended to determine the type of unintentional non-adherence.

IPD SHARING:
Plan to Share IPD: No
The information will be anonymized by the Principal Investigator (PI)

REFERENCES:
- [Background] Frey SM, Fagnano M, Halterman JS. Adolescent Knowledge of When to Use Inhaled Asthma Medications: Implications for Management. J Adolesc Health. 2023 Apr;72(4):623-628. doi: 10.1016/j.jadohealth.2022.10.034. Epub 2022 Dec 15. PMID 36528520
- [Background] Manti S, Licari A, Leonardi S, Marseglia GL. Management of asthma exacerbations in the paediatric population: a systematic review. Eur Respir Rev. 2021 Jul 13;30(161):200367. doi: 10.1183/16000617.0367-2020. Print 2021 Sep 30. PMID 34261742
- [Background] Kosse RC, Koster ES, Kaptein AA, de Vries TW, Bouvy ML. Asthma control and quality of life in adolescents: The role of illness perceptions, medication beliefs, and adherence. J Asthma. 2020 Oct;57(10):1145-1154. doi: 10.1080/02770903.2019.1635153. Epub 2019 Jul 5. PMID 31225980
- [Background] Ciprandi G, Licari A, Castagnoli R, Ciprandi R, Marseglia GL. Asthma control in adolescents: the importance of assessing adherence. Acta Biomed. 2022 Aug 31;93(4):e2022264. doi: 10.23750/abm.v93i4.12448. PMID 36043978
- [Background] Lizano-Barrantes C, Garin O, Mayoral K, Dima AL, Pont A, Caballero-Rabasco MA, Praena-Crespo M, Valdesoiro-Navarrete L, Guerra MT, Bercedo-Sanz A, Ferrer M. Impact of treatment adherence and inhalation technique on asthma outcomes of pediatric patients: a longitudinal study. Front Pharmacol. 2024 Mar 13;15:1340255. doi: 10.3389/fphar.2024.1340255. eCollection 2024. PMID 38549668
- [Background] Basharat S, Jabeen U, Zeeshan F, Bano I, Bari A, Rathore AW. Adherence to asthma treatment and their association with asthma control in children. J Pak Med Assoc. 2018 May;68(5):725-728. PMID 29885170
- [Background] McCrossan P, Shields MD, McElnay JC. Medication Adherence in Children with Asthma. Patient Prefer Adherence. 2024 Mar 5;18:555-564. doi: 10.2147/PPA.S445534. eCollection 2024. PMID 38476591
- [Background] Gonzalez Betlza M, Bruno I, Yemini L, Zuniga C, Bello Pedrosa O. [Impact of a program of health education for the asthmatic child and their families]. Arch Argent Pediatr. 2020 Apr;118(2):145-149. doi: 10.5546/aap.2020.145. Spanish. PMID 32199068
- [Background] Capanoglu M, Dibek Misirlioglu E, Toyran M, Civelek E, Kocabas CN. Evaluation of inhaler technique, adherence to therapy and their effect on disease control among children with asthma using metered dose or dry powder inhalers. J Asthma. 2015 Oct;52(8):838-45. doi: 10.3109/02770903.2015.1028075. Epub 2015 Jun 2. PMID 26037396
- [Background] Almomani BA, Al-Qawasmeh BS, Al-Shatnawi SF, Awad S, Alzoubi SA. Predictors of proper inhaler technique and asthma control in pediatric patients with asthma. Pediatr Pulmonol. 2021 May;56(5):866-874. doi: 10.1002/ppul.25263. Epub 2021 Jan 26. PMID 33497530
- [Background] Tao S, Fan Q, Hariharan VS, Zhi H. Effectiveness of nursing interventions for management of children with bronchial asthma: A systematic review and meta-analysis. Int J Nurs Pract. 2023 Dec;29(6):e13139. doi: 10.1111/ijn.13139. Epub 2023 Mar 6. PMID 36879363
- [Background] Normansell R, Kew KM, Mathioudakis AG. Interventions to improve inhaler technique for people with asthma. Cochrane Database Syst Rev. 2017 Mar 13;3(3):CD012286. doi: 10.1002/14651858.CD012286.pub2. PMID 28288272
- [Background] Roche N, Aggarwal B, Boucot I, Mittal L, Martin A, Chrystyn H. The impact of inhaler technique on clinical outcomes in adolescents and adults with asthma: A systematic review. Respir Med. 2022 Oct;202:106949. doi: 10.1016/j.rmed.2022.106949. Epub 2022 Sep 2. PMID 36063773
- [Background] Sanchis J, Gich I, Pedersen S; Aerosol Drug Management Improvement Team (ADMIT). Systematic Review of Errors in Inhaler Use: Has Patient Technique Improved Over Time? Chest. 2016 Aug;150(2):394-406. doi: 10.1016/j.chest.2016.03.041. Epub 2016 Apr 7. PMID 27060726
- [Background] Price DB, Roman-Rodriguez M, McQueen RB, Bosnic-Anticevich S, Carter V, Gruffydd-Jones K, Haughney J, Henrichsen S, Hutton C, Infantino A, Lavorini F, Law LM, Lisspers K, Papi A, Ryan D, Stallberg B, van der Molen T, Chrystyn H. Inhaler Errors in the CRITIKAL Study: Type, Frequency, and Association with Asthma Outcomes. J Allergy Clin Immunol Pract. 2017 Jul-Aug;5(4):1071-1081.e9. doi: 10.1016/j.jaip.2017.01.004. Epub 2017 Mar 9. PMID 28286157
- [Background] Moral Gil L, Asensi Monzó M, Juliá Benito JC, Ortega Casanueva C, Paniagua Calzón NM, Pérez García MI, Rodríguez Fernández-Oliva CR, Sanz Ortega J, Valdesoiro Navarrete L, Valverde Molina J. Asma en pediatría. Consenso regAp. Alicante (España): Luis Morales; 2021. Disponible en: https://neumoped.org/wp-content/uploads/2021/02/Asma-en-pediatria-consenso-regap-2021_94549.pdf

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT07364643/Prot_SAP_000.pdf
  • Informed Consent Form: Participant consent for children aged 6-10 years (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT07364643/ICF_001.pdf
  • Informed Consent Form: Participant consent for children aged 11-17 years (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT07364643/ICF_002.pdf